CLINICAL TRIAL: NCT00254631
Title: Preemptive Analgesia With OxyContin Versus Placebo Before Surgery for Long Bone Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, edery, Rambam Health Care Campus, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pre-oxy.CTIL
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Fractures
Keywords: long bone fracture; open fractures; closed fractures; trauma
MeSH Terms: conditions — Fractures, Bone; Fractures, Open; Fractures, Closed; Wounds and Injuries | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- study group (Active Comparator): pre operative medication with 20 mg oxycontine PO
  Interventions: Drug: Oxycodone hydrochloride
- placebo group (Placebo Comparator): pre operative medication with placebo tablet PO

INTERVENTIONS:
Drug: Oxycodone hydrochloride
  Arms: study group

SUMMARY:
We would like to check whether pre-operative administration of an oral controlled-release opioid formulation (Oxycodone hydrochloride (OxyContin)) could result in a clear effect of preemptive analgesia.

DETAILED DESCRIPTION:
Preemptive analgesia is based on the concept of treating pain before inflicting the painful stimulus. One suggested mechanism is that transmission of pain signals is altered when the patient is treated before infliction of noxious stimulation. That prevents changes from happening in the nervous system, making transformation from acute to chronic pain ("central sensitization") less likely, and thus reducing post operative pain.

Clinically, good post operative pain control has been shown to be an effective method for hastening patient convalescence and discharge. It makes part of a general approach aiming to accelerate surgical recovery through earlier enteric feeding and ambulation

OxyContin tablets deliver Oxycodone at a controlled release manner, over 12 hours. After oral administration oral bioavailability is 60-87%.

A biphasic absorption pattern is observed, describing the initial (0.6 hours) and prolonged (6.9 hours) release of Oxycodone from the OxyContin tablets. Clinical analgesia is observed within 1 hour of administration.

We believe that this mode of oral drug release is more appropriate for the perioperative pain treatment of patients undergoing short to medium term operations: with timely administration, the first absorbed part of the drug reaches the plasma before infliction of the noxious stimuli, possibly counteracting primary sensitization, and the second part absorbed, acts on post operative ongoing pain, possibly counteracting more advanced stages of neuronal plasticity.

Study Hypothesis:

Our hypothesis is that post operative pain will be lowered by pre-operative administration of OxyContin. When comparing the two groups we will look for differences in observed parameters, especially VAS numbers, time to first analgesic request, post operative analgesic requirements, time to first oral intake and length of hospitalization, to confirm or deny our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consent.
2. Age 18 years to 60 years.
3. Isolated limb bone fracture/s.

Exclusion Criteria:

1. Patient refusal.
2. Age 61 years and older.
3. Known allergy to study medication.
4. Multiple bone fractures in different limbs.
5. Multiple trauma.
6. Oncological patients.
7. Respiratory depression / respiratory insufficiency / hypercarbia.
8. Acute bronchial asthma.
9. CNS depression / hallucinations.
10. Alzheimer / dementia.
11. Known convulsive disorder.
12. Prostate hypertrophy.
13. Paralytic ileus.
14. Renal dysfunction (plasma creatinine > 1.5).
15. Liver dysfunction.
16. Adrenocortical insufficiency.
17. Hypothyroidism.
18. Pancreatitis.
19. Pregnancy and lactating.
20. Drug abuse, current or in the past.
21. Alcohol abuse on admission to operating room.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
post operative pain scores during first 24 hours (Visual analog scale) | 24 hours after surgery

SECONDARY OUTCOMES:
Time to first analgesic request | at PACU
Total other pain medications at first 24 hours post operative | first 24 hours after surgery
Time to first oral intake | first 24 hours after surgery
Length of hospitalization | after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Edery, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- RAMBAM Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Bach S, Noreng MF, Tjellden NU. Phantom limb pain in amputees during the first 12 months following limb amputation, after preoperative lumbar epidural blockade. Pain. 1988 Jun;33(3):297-301. doi: 10.1016/0304-3959(88)90288-6. PMID 3419837
- [Background] Code WE, Yip RW, Rooney ME, Browne PM, Hertz T. Preoperative naproxen sodium reduces postoperative pain following arthroscopic knee surgery. Can J Anaesth. 1994 Feb;41(2):98-101. doi: 10.1007/BF03009799. PMID 8131242
- [Background] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Ong CK, Lirk P, Seymour RA, Jenkins BJ. The efficacy of preemptive analgesia for acute postoperative pain management: a meta-analysis. Anesth Analg. 2005 Mar;100(3):757-773. doi: 10.1213/01.ANE.0000144428.98767.0E. PMID 15728066